CLINICAL TRIAL: NCT00791297
Title: A Phase 2, Randomized Study to Evaluate the Safety and Efficacy of Two Contraceptive Vaginal Rings Delivering a Daily Dose of 1500 or 2500 μg of CDB-2914 on Inhibition of Ovulation, Endometrial Changes and Bleeding Patterns in Normal Cycling Women
Brief Title: Study to Evaluate the Safety and Efficacy of Two Contraceptive Vaginal Rings Delivering a Daily Dose of 1500 or 2500 μg of CDB-2914
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Population Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Population Council #422
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Contraception
Keywords: CDB-2914; Contraceptive Vaginal Rings; ovulation; endometrial changes; bleeding patterns; normal cycling women; Inhibition of ovulation, endometrial changes and bleeding patterns in normal cycling women
MeSH Terms: interventions — ulipristal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Contraceptive Vaginal Ring delivering a daily dose of 1500 μg of CDB-2914
  Interventions: Drug: CDB-2914
- 2 (Active Comparator): Contraceptive Vaginal Ring delivering a daily dose of 2500 μg of CDB-2914
  Interventions: Drug: CDB-2914

INTERVENTIONS:
Drug: CDB-2914 — Contraceptive Vaginal Rings delivering a daily dose of 1500 or 2500 μg of CDB-2914

SUMMARY:
The purpose of this study is to to determine pharmacodynamic effects of a vaginal ring delivering either 1,500 or 2,500 μg of CDB-2914 per day during 6 months of treatment on:

1. follicular function and inhibition of ovulation
2. the endometrium
3. bleeding patterns; and also to assess safety including effects on the endometrium

ELIGIBILITY:
Inclusion Criteria:

* Healthy women of reproductive age (21-40 years)
* Not at risk for pregnancy based on one of the following
* subject has undergone sterilization
* subject is monogamous and her male partner has undergone sterilization
* subject agrees to be abstinent for the entire duration of the study (Oregon site only)
* subject does not have sex with men (Oregon site only)
* Have regular menstrual cycles of 25-35 days duration
* Have an intact uterus and both ovaries
* Will be able to comply with the protocol
* Capable of giving informed consent

Exclusion Criteria:

* Women participating in another clinical trial
* Women not living in the catchment area of the clinic
* Known hypersensitivity to progestins or antiprogestins
* Known hypersensitivity to silicone rubber
* Any chronic disease
* All contraindications to oral contraceptive use, including
* Thrombophlebitis or thromboembolic disorders
* Past history of deep vein thrombophlebitis or thromboembolic disorders
* Past or current cerebrovascular or coronary artery disease
* Migraine with focal aura
* Known or suspected carcinoma of the breast
* Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia
* Undiagnosed abnormal genital bleeding
* Cholestatic jaundice of pregnancy or jaundice with prior pill use
* Hepatic adenomas or carcinomas
* Known or suspected pregnancy
* Desire to get pregnant during the study (through the use of reproductive technology for sterilized women or vasectomy reversal for sterilized partners)
* Breastfeeding
* Undiagnosed vaginal discharge or vaginal lesions or abnormalities
* Elevated Prolactin levels (above laboratory normal values)
* Women with a current abnormal Pap
* In accordance with the Bethesda system of classification smear suggestive of high-grade pre-cancerous lesion(s), including HGSIL, are excluded
* Women with LGSIL or ASCUS/high-risk HPV positive may participate if further evaluated with colposcopy and biopsy and no evidence of a lesion with a severity > CIN I is present and/or endocervical curettage is negative
* Women with a biopsy finding of CIN I should have follow up for this finding per standard of care; women are excluded it treatment is indicated
* In accordance with other Pap class systems
* Women with high grade dysplasia are excluded
* Women with low grade dysplasia or CIN I interpretation on Pap smear may participate based on Investigator discretion and provided there is appropriate follow up in accordance with local standards of care
* Known benign or malignant liver tumors; known active liver disease
* Cancer (past history of any carcinoma or sarcoma)
* Medically diagnosed severe depression currently or in the past
* Known or suspected alcoholism or drug abuse
* Abnormal serum fasting clinical chemistry values
* Women with known abnormal thyroid status
* Women with known impaired hypothalamic-pituitary-adrenal reserve
* Average diastolic BP > 85 mm or systolic BP >135 mm Hg after 5-10 minutes rest
* Body mass index(BMI) > 29.0
* Smoking in women who are 35 years and over or will be 35 years during the course of the trial; women < 35 years who smoke greater than 15 cigarettes per day must be evaluated by the PI for inclusion based on risk factors that would increase their risk for CVD and thromboembolism, e.g. lipid levels, glucose level, BP, BMI, family history of CVD at a young age
* Women with severe cystoceles or rectoceles
* Use within the past 2 months of any implanted hormonal contraceptives including Mirena [progestin containing intrauterine system (IUS)] or Norplant (subdermal implant delivering LNG) NOTE: Removal of implanted hormonal contraceptives must have been for personal reasons unrelated to the purpose of enrollment in this study
* Current use of a non-hormone containing IUD. NOTE: Removal of an IUD must have been for personal reasons unrelated to the purpose of enrollment in this study
* Use of injectable contraceptives during the previous 3 months (e.g. Cyclofem) or 6 months (e.g. DMPA)
* Women who do not have at least two progesterone measurements during the control cycle of ≥10nmol/L will be excluded from further participation in the study (See Section 13.41)

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2008-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable will be ovulation suppression measured by progesterone serum levels. | All women will use the assigned CVR for 6 months

SECONDARY OUTCOMES:
Regular follow-up of follicle diameter will be made with USS to determine the timing of ovulation or, in the absence of ovulation, the fate of the dominant follicle. | All women will use the assigned CVR for 6 months
Clinical safety will be evaluated and the effects on the endometrium will be measured. | All women will use the assigned CVR for 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- Oregon Health & Science University, Portland, Oregon, United States
- Instituto Chileno de Medicina Reproductiva, Santiago, Chile
- Profamilia, Santo Domingo, Dominican Republic